CLINICAL TRIAL: NCT04221113
Title: Principle Investigator
Brief Title: Functional Recovery Measurement : Comparing Early Active Mobilization Versus Immobilization After Extensor Tendon Repair in Zones IV to VIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Zaara Zahid, Principle investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1365
Record Dates: First submitted 2019-12-16; First posted 2020-01-09 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Injury of Extensor Tendon of Hand (Disorder)
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Healthy patients with only extensor tendon injuries will be recruited in this study and will randomly divided in two groups. An intervention in the form of rehabilitation will be given to patients in two different protocols than outcomes will be assessed.
Who Masked: Participant
Masking Description: This study will be single blinded means that patient will be unaware of protocol written inside the envolupe.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A ( Immobilization protocol) (Active Comparator): Group A patients will receive static splints.By the end of 4 weeks the splint will be modified and patients will start doing physiotherapy. Movement at MCPJ will be from 0 to 45 degrees.
  Interventions: Procedure: physiotherapy
- Group B( early active mobilization protocol). (Active Comparator): Group B patients will receive splints in such a way that from 3rd post operative day patients will be instructed to do physiotherapy. Initially MCPJ movement will be from 0 to 30 degrees.
  Interventions: Procedure: physiotherapy

INTERVENTIONS:
Procedure: physiotherapy — Two protocols have been described for physiotherapy of post extensor tendon injuries. one is immobilization till 3 weeks and than gradual increase in active motion of hand. The second protocol is early active motion. this would be done under senior physiotherapist.

SUMMARY:
Functional recovery measurement : Comparing early active mobilization versus immobilization after extensor tendon repair in zones IV to VIII.

Immobilization for six weeks has been the postoperative protocol for the patients with hand's extensor tendon repair in our institute. In this study early mobilization of the hand i.e. also an internationally followed way, is compared with the aforementioned immobilization protocol to see which turns out to be a better option in the interest of the patient.

DETAILED DESCRIPTION:
patients selection in both groups will be random by using close envolupe technique.

In group A ( immobilisation) physiotherapy will start by the end of 4th week and the upper limit of flexion would be 45 degrees.

In group B ( EAM) physiotherapy will start by the end of 1st week and the upper limit of flexion would be 30 degrees.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender having simple lacerations of extrinsic extensor tendons · of the hand in · Verdan's zones IV-VIII

  * Age range 18 to 65 years
  * Sharp Cut Injury

Exclusion Criteria:

* Patients with complex injured hands like significant skin loss, bone and/or joint injuries. · Flexor tendon injuries.

  * Partial tendon lacerations
  * Tendon injuries at multiple levels

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
To measure total active motion in the results of both groups to compare which one has better results. | 8 weeks
  Flexion range and extension lag at each joint i.e MCPJ, PIPJ and DIPJ will be assessed at 2, 4 and 8 weeks of follow up. By using this following formula total active motion at each joint mentioned above will be assessed.
  TAM is calculated by the following formula:
  TAM =([MCPJ +PIPJ +DIPJ flexion]- [MCPJ +PIPJ +DIPJ extension lag

CONTACTS AND LOCATIONS:
Locations (1):
- Zaara Zahid, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sameem M, Wood T, Ignacy T, Thoma A, Strumas N. A systematic review of rehabilitation protocols after surgical repair of the extensor tendons in zones V-VIII of the hand. J Hand Ther. 2011 Oct-Dec;24(4):365-72; quiz 373. doi: 10.1016/j.jht.2011.06.005. Epub 2011 Sep 1. PMID 21889303
- See also: To determine which rehabilitation protocol yields the best outcomes with respect to range of motion and grip strength in extensor zones V-VIII of the hand — https://www.ncbi.nlm.nih.gov/pubmed/21889303